CLINICAL TRIAL: NCT02547623
Title: A Phase 3, Prospective, Randomized, Parallel-design, Multicenter Study to Evaluate the Safety of Icon Bioscience-10090 for the Treatment of Inflammation Associated With Cataract Surgery
Brief Title: Study to Evaluate the Safety for the Treatment of Inflammation Associated With Cataract Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ICON Bioscience Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C15-01
Record Dates: First submitted 2015-09-09; First posted 2015-09-11 (Estimated); Results first posted 2018-06-19 (Actual); Last update posted 2018-08-21 (Actual); Status verified 2018-07

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract | interventions — Dexamethasone; Calcium Dobesilate; Prednisolone; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- dexamethasone depot (Active Comparator): dexamethasone depot 517 mcg
  Interventions: Drug: Dexamethasone
- standard of care (Active Comparator): prednisolone drops 1%
  Interventions: Drug: Prednisolone

INTERVENTIONS:
Drug: Dexamethasone — depot intracameral
  Other Names: Dexycu
  Arms: dexamethasone depot
Drug: Prednisolone — Prednisolone eye drops 1%
  Other Names: standard of care
  Arms: standard of care

SUMMARY:
The study is a prospective, randomized, parallel-design, multicenter trial in patients ≥40 years of age undergoing cataract surgery. Patients who meet all inclusion and no exclusion criteria will be randomized to 1 of 2 treatment groups

* A single 5 mcl anterior chamber injection of IBI 10090, 103.4 mcg/mcl dexamethasone, equivalent dexamethasone dose: 517 mcg at the conclusion of cataract surgery or;
* Prednisolone acetate ophthalmic suspension 1% eye drops administered 1 drop 4 times daily (QID) for 3 weeks Safety will be assessed by adverse events (AEs), slit lamp biomicroscopy, fundus examination, intraocular pressure (IOP), visual acuity, and specular microscopy endothelial cell count.

DETAILED DESCRIPTION:
The study is a prospective, randomized, parallel-design, multicenter trial in patients ≥40 years of age undergoing cataract surgery. Patients who meet all inclusion and no exclusion criteria will be randomized to 1 of 2 treatment groups

* A single 5 mcl anterior chamber injection of IBI 10090, 103.4 mcg/mcl dexamethasone, equivalent dexamethasone dose: 517 mcg at the conclusion of cataract surgery or;
* Prednisolone acetate ophthalmic suspension 1% eye drops administered 1 drop 4 times daily (QID) for 3 weeks

ELIGIBILITY:
Inclusion Criteria:

* undergoing cataract surgery

Exclusion Criteria:

* glaucoma patient, pregnancy, allergy to dexamethasone

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2015-11-06 (Actual); Primary Completion 2016-08-16 (Actual); Study Completion 2016-08-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Donnenfeld, MD, Principal Investigator — Ophthalmic Consultants of Long Island
Locations (11):
- United States (11):
  - Kislinger MD inc, Glendora, California
  - Inland Eye Specialists, Hemet, California
  - Harvard Eye Associated, Laguna Hills, California
  - Feinerman Vision Center, Newport Beach, California
  - Cincinnati Eye Institute, Edgewood, Kentucky
  - Associated Eye Care, Stillwater, Minnesota
  - Matossian Eye Associates, Pennington, New Jersey
  - Ophthalmic Consultants of Long Island, Garden City, New York
  - Cincinnati Eye Institute, Cincinnati, Ohio
  - Carolina Eye Care Physicians, Mt. Pleasant, South Carolina
  - the eye institute of Utah, Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first patient was enrolled into the study on 06 November 2015 and the last patient completed the study on 16 August 2016.
Pre-assignment Details: Of the 194 patients randomized, 181 patients were dosed and included in the ITT (intent-to-treat) and safety analysis sets. 13 randomized patients were not dosed and terminated from the study. Some of the patients that were not dosed had at least one significant protocol deviation.
Groups:
- Dexamethasone Depot: A single intraocular dose of dexamethasone (517 mcg) at the conclusion of cataract surgery
- Prednisolone Drops 1% (Standard of Care): Three weeks of treatment with prednisolone drops 1% (one drop, four times daily for three weeks)
Period: Overall Study
Arm/Group | Dexamethasone Depot | Prednisolone Drops 1% (Standard of Care)
Started | 126 | 55
Completed | 122 | 52
Not Completed | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dexamethasone Depot | Prednisolone Drops 1% (Standard of Care) | Total
Number analyzed (Participants) | 126 | 55 | 181
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 34 | 17 | 51
  >=65 years | 92 | 38 | 130
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 31 | 98
  Male | 59 | 24 | 83
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 1 | 10
  Not Hispanic or Latino | 117 | 54 | 171
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 1 | 12
  White | 111 | 52 | 163
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 0 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 126 | 55 | 181
Study Eye [Number; unit: study eye]
  OD (Right eye) | 67 | 27 | 94
  OS (Left eye) | 59 | 28 | 87
Best Corrected Visual Acuity [Mean (Standard Deviation); unit: LogMar] — Visual Acuity assessed by the Snellen chart, was expressed as the logarithm of the minimum angle of resolution (logMAR), and could range from 0 (representing 20/20 vision) to 1
  LogMar
    study eye number | .292 (.1913) | .355 (.2557) | .311 (.2141)
    fellow eye number | .126 (.1394) | .176 (.2123) | .141 (.1660)
Corneal Endothelial Cell Density - Specular Microscopy [Mean (Standard Deviation); unit: cells/mm^2] | 2491.91 (346.365) | 2398.33 (384.092) | 2463.15 (359.902)
Intraocular Pressure [Mean (Standard Deviation); unit: mmHg]
  Study eye | 15.1 (2.94) | 14.4 (2.71) | 14.9 (2.88)
  Fellow eye | 14.9 (2.88) | 14.5 (2.79) | 14.8 (2.85)
Use of Viscoelastic during the Surgery [Count of Participants; unit: Participants]
  Yes | 126 | 55 | 181
  No | 0 | 0 | 0
Use of Femto prior to the Surgery [Count of Participants; unit: Participants]
  Yes | 25 | 8 | 33
  No | 101 | 47 | 148

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: Treatment-emergent Adverse Events were defined as events that started after the study drug administration, and occurred before termination of the study, or were present before study drug administration and worsened after dose administration.
Time Frame: Baseline to postoperative day 90/ early termination
Measure: Count of Participants; unit: Participants
Arm/Group | Dexamethasone Depot | Prednisolone Drops 1% (Standard of Care)
Number analyzed (Participants) | 126 | 55
Participants
  Ocular events: study eye: Any TEAE | 53 | 13
  Ocular events: study eye: Serious TEAE | 1 | 0
  Ocular events: study eye: No TEAE | 72 | 42
  Ocular events: fellow eye: Any TEAE | 12 | 4
  Ocular events: fellow eye: Serious TEAE | 0 | 0
  Ocular events: fellow eye: No TEAE | 114 | 51
  Systemic events: Any TEAE | 10 | 6
  Systemic events: Serious TEAE | 2 | 0
  Systemic events: No TEAE | 114 | 49

2. Secondary Outcome: Intraocular Pressure Measurement
Description: Intraocular Pressure was measured by Goldmann applanation tonometry.
Time Frame: Baseline, Postoperative (POD) 1, POD 8, POD 30, POD 90/Early termination
Measure: Mean (Standard Deviation); unit: mmHG
Arm/Group | Dexamethasone Depot | Prednisolone Drops 1% (Standard of Care)
Number analyzed (Participants) | 126 | 55
mmHG
  Screening (Baseline) | 15.1 (2.94) | 14.4 (2.71)
  Post Operative Day 1 | 19.1 (6.54) | 17.5 (6.44)
  Post Operative Day 8 | 15.0 (4.7) | 15.1 (3.64)
  Post Operative Day 30 | 13.8 (3.2) | 14.1 (3.57)
  Post Operative Day 90/End of Treatment | 13.0 (2.89) | 12.7 (2.93)

3. Secondary Outcome: Visual Acuity in Study Eye
Description: Visual Acuity assessed by the Snellen chart, was expressed as the logarithm of the minimum angle of resolution (logMAR), and could range from 0 (representing 20/20 vision) to 1
Time Frame: Baseline, Postoperative (POD) 1, POD 8, POD 30, POD 90/Early termination
Measure: Mean (Standard Deviation); unit: LogMar
Arm/Group | Dexamethasone Depot | Prednisolone Drops 1% (Standard of Care)
Number analyzed (Participants) | 126 | 55
LogMar
  Screening (Baseline) | .292 (0.1913) | .355 (.2557)
  Post Operative Day 1 | .249 (.1398) | .327 (.2129)
  Post Operative Day 8 | .073 (.1353) | .073 (.1746)
  Post Operative Day 30 | .039 (.0952) | .040 (.1350)
  Post Operative Day 90/End of Treatment | .040 (.1012) | .047 (.1150)

4. Secondary Outcome: Slit Lamp Biomicroscopy - Conjunctival Hyperemia Grade
Description: Slit lamp biomicroscopy of the anterior chamber was performed using a slit beam of 1-mm height and 1-mm width with maximum luminance through the highest-powered lens using the Investigator's standard slit lamp equipment and procedure.
  Conjunctiva hyperemia slit lamp results were summarized by treatment group and time point.
Time Frame: Baseline, Postoperative (POD) 1, POD 8, POD 30, POD 90/Early termination
Measure: Count of Participants; unit: Participants
Arm/Group | Dexamethasone Depot | Prednisolone Drops 1% (Standard of Care)
Number analyzed (Participants) | 126 | 55
Participants
  Baseline: 0 (Absent) | 124 | 55
  Baseline: 1 (Mild) | 1 | 0
  Baseline: 2 (Moderate) | 1 | 0
  Baseline: 3 (Severe) | 0 | 0
  Baseline: No value | 0 | 0
  Postoperative day 1: 0 (Absent) | 103 | 45
  Postoperative day 1: 1 (Mild) | 21 | 10
  Postoperative day 1: 2 (Moderate) | 2 | 0
  Postoperative day 1: 3 (Severe) | 0 | 0
  Postoperative day 1: No value | 0 | 0
  Postoperative day 8: 0 (Absent) | 115 | 45
  Postoperative day 8: 1 (Mild) | 11 | 8
  Postoperative day 8: 2 (Moderate) | 0 | 0
  Postoperative day 8: 3 (Severe) | 0 | 0
  Postoperative day 8: No value | 0 | 2
  Postoperative day 30: 0 (Absent) | 107 | 44
  Postoperative day 30: 1 (Mild) | 14 | 8
  Postoperative day 30: 2 (Moderate) | 2 | 0
  Postoperative day 30: 3 (Severe) | 0 | 0
  Postoperative day 30: No value | 3 | 3
  Postoperative day 90/End of Treatment: 0 (Absent) | 119 | 50
  Postoperative day 90/End of Treatment: 1 (Mild) | 4 | 2
  Postoperative day 90/End of Treatment: 2 (Moderate) | 0 | 0
  Postoperative day 90/End of Treatment: 3 (Severe) | 0 | 0
  Postoperative day 90/End of Treatment: No value | 3 | 3

5. Secondary Outcome: Slit Lamp Biomicroscopy - Cornea Edema Grade
Description: Slit lamp biomicroscopy of the anterior chamber was performed using a slit beam of 1-mm height and 1-mm width with maximum luminance through the highest-powered lens using the Investigator's standard slit lamp equipment and procedure.
  Cornea edema slit lamp results in the study eye were summarized by treatment group and time point.
Time Frame: Baseline, Postoperative (POD) 1, POD 8, POD 30, POD 90/Early termination
Measure: Count of Participants; unit: Participants
Arm/Group | Dexamethasone Depot | Prednisolone Drops 1% (Standard of Care)
Number analyzed (Participants) | 126 | 55
Participants
  Baseline: 0 (Absent) | 126 | 54
  Baseline: 1 (Mild) | 0 | 0
  Baseline: 2 (Moderate) | 0 | 0
  Baseline: 3 (Severe) | 0 | 0
  Baseline: No value | 0 | 1
  Postoperative day 1: 0 (Absent) | 74 | 37
  Postoperative day 1: 1 (Mild) | 43 | 15
  Postoperative day 1: 2 (Moderate) | 9 | 3
  Postoperative day 1: 3 (Severe) | 0 | 0
  Postoperative day 1: No value | 0 | 0
  Postoperative day 8: 0 (Absent) | 109 | 48
  Postoperative day 8: 1 (Mild) | 16 | 6
  Postoperative day 8: 2 (Moderate) | 0 | 0
  Postoperative day 8: 3 (Severe) | 0 | 0
  Postoperative day 8: No value | 1 | 1
  Postoperative day 30: 0 (Absent) | 121 | 52
  Postoperative day 30: 1 (Mild) | 0 | 0
  Postoperative day 30: 2 (Moderate) | 2 | 0
  Postoperative day 30: 3 (Severe) | 0 | 0
  Postoperative day 30: No value | 3 | 3
  Postoperative day 90/End of Treatment: 0 (Absent) | 123 | 52
  Postoperative day 90/End of Treatment: 1 (Mild) | 0 | 0
  Postoperative day 90/End of Treatment: 2 (Moderate) | 0 | 0
  Postoperative day 90/End of Treatment: 3 (Severe) | 0 | 0
  Postoperative day 90/End of Treatment: No value | 3 | 3

6. Secondary Outcome: Summary of Concomitant Medications Used in the Study Eye or Both Eyes
Time Frame: Baseline, Postoperative (POD) 1, POD 8, POD 30, POD 90/Early termination
Measure: Count of Participants; unit: Participants
Arm/Group | Dexamethasone Depot | Prednisolone Drops 1% (Standard of Care)
Number analyzed (Participants) | 126 | 55
Participants
  Patients reporting at least one concomitant medica | 124 | 55
  Antiseptics and disinfectants | 1 | 1
  Anesthetics | 4 | 1
  Psycholeptics | 2 | 1
  Ophthalmologicals | 124 | 55
  Thyroid therapy | 0 | 1

7. Secondary Outcome: Changes in the Corneal Endothelial Cell Count
Description: Corneal Endothelial Cell Density was measured by specular microscopy.
Time Frame: Baseline, Postoperative day 90/Early termination
Measure: Mean (Standard Deviation); unit: cells/mm^2
Arm/Group | Dexamethasone Depot | Prednisolone Drops 1% (Standard of Care)
Number analyzed (Participants) | 126 | 55
cells/mm^2
  Baseline | 2483.66 (351.819) | 2398.33 (384.092)
  Postoperative day 90/End of treatment | 2141.77 (522.327) | 2106.39 (517.938)
  Change from Baseline | -334.60 (415.071) | -288.83 (376.775)

8. Secondary Outcome: Optic Disc Cup-disc Ratio for the Study Eye
Description: Calculated as the ratio of the diameter of the depression (cup) to that of the optical nerve head (disc).
Time Frame: Baseline, POD 90/Early termination
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Dexamethasone Depot | Prednisolone Drops 1% (Standard of Care)
Number analyzed (Participants) | 126 | 55
ratio
  Screening (Baseline) | .31 (.142) | .32 (.135)
  Postoperative day 90/End of treatment | .31 (.131) | .33 (.143)

9. Secondary Outcome: Dilated Opthalmoscopy Findings - Optic Disc (Study Eye)
Description: The number and percentage of patients with normal or abnormal findings from dilated opthalmoscopy examination of the study eye's optic disc
Time Frame: Baseline, POD 90/Early termination
Measure: Count of Participants; unit: Participants
Arm/Group | Dexamethasone Depot | Prednisolone Drops 1% (Standard of Care)
Number analyzed (Participants) | 126 | 55
Participants
  Screening (Baseline): Normal | 115 | 52
  Screening (Baseline): Abnormal | 2 | 1
  Screening (Baseline): Not analyzed | 9 | 2
  Postoperative day 90/End of treatment: Normal | 119 | 50
  Postoperative day 90/End of treatment: Abnormal | 2 | 1
  Postoperative day 90/End of treatment: Not analyzed | 5 | 4

10. Secondary Outcome: Dilated Opthalmoscopy Findings - Retina (Study Eye)
Description: The number and percentage of patients with normal or abnormal findings from dilated opthalmoscopy examination of the study eye's retina
Time Frame: Baseline, POD 90/Early termination
Measure: Count of Participants; unit: Participants
Arm/Group | Dexamethasone Depot | Prednisolone Drops 1% (Standard of Care)
Number analyzed (Participants) | 126 | 55
Participants
  Screening (Baseline): Normal | 120 | 51
  Screening (Baseline): Abnormal | 5 | 4
  Screening (Baseline): Not analyzed | 1 | 0
  Postoperative day 90/End of treatment: Normal | 118 | 50
  Postoperative day 90/End of treatment: Abnormal | 5 | 1
  Postoperative day 90/End of treatment: Not analyzed | 3 | 4

11. Secondary Outcome: Dilated Opthalmoscopy Findings - Macula (Study Eye)
Description: The number and percentage of patients with normal or abnormal findings from dilated opthalmoscopy examination of the study eye's macula.
Time Frame: Baseline, POD 90/Early termination
Measure: Count of Participants; unit: Participants
Arm/Group | Dexamethasone Depot | Prednisolone Drops 1% (Standard of Care)
Number analyzed (Participants) | 126 | 55
Participants
  Screening (Baseline): Normal | 109 | 44
  Screening (Baseline): Abnormal | 15 | 11
  Screening (Baseline): Not analyzed | 2 | 0
  Postoperative day 90/End of treatment: Normal | 107 | 39
  Postoperative day 90/End of treatment: Abnormal | 16 | 12
  Postoperative day 90/End of treatment: Not analyzed | 3 | 4

12. Secondary Outcome: Dilated Opthalmoscopy Findings - Choroid (Study Eye)
Description: The number and percentage of patients with normal or abnormal findings from dilated opthalmoscopy examination of the study eye's choroid
Time Frame: Baseline, POD 90/Early termination
Measure: Count of Participants; unit: Participants
Arm/Group | Dexamethasone Depot | Prednisolone Drops 1% (Standard of Care)
Number analyzed (Participants) | 126 | 55
Participants
  Screening (Baseline): Normal | 124 | 54
  Screening (Baseline): Abnormal | 0 | 0
  Screening (Baseline): Not analyzed | 2 | 1
  Postoperative day 90/End of treatment: Normal | 122 | 50
  Postoperative day 90/End of treatment: Abnormal | 1 | 0
  Postoperative day 90/End of treatment: Not analyzed | 3 | 5

13. Secondary Outcome: Dilated Opthalmoscopy Findings - Vitreous (Study Eye)
Description: The number and percentage of patients with normal or abnormal findings from dilated opthalmoscopy examination of the study eye's vitreous
Time Frame: Baseline, POD 90/Early termination
Measure: Count of Participants; unit: Participants
Arm/Group | Dexamethasone Depot | Prednisolone Drops 1% (Standard of Care)
Number analyzed (Participants) | 126 | 55
Participants
  Screening (Baseline): Normal | 104 | 49
  Screening (Baseline): Abnormal | 21 | 5
  Screening (Baseline): Not analyzed | 1 | 1
  Postoperative day 90/End of treatment: Normal | 107 | 44
  Postoperative day 90/End of treatment: Abnormal | 16 | 7
  Postoperative day 90/End of treatment: Not analyzed | 3 | 4

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from screening until postoperative day 90/end of treatment.
Arm/Group | Dexamethasone Depot | Prednisolone Drops 1% (Standard of Care)
All-Cause Mortality (participants affected / at risk) | 0/126 | 0/55
Serious Adverse Events (participants affected / at risk) | 3/126 | 0/55
Other Adverse Events (participants affected / at risk) | 23/126 | 6/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dexamethasone Depot (N=126) | Prednisolone Drops 1% (Standard of Care) (N=55)
Diabetic retinopathy (Eye disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0
Abdominal hernia (Gastrointestinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dexamethasone Depot (N=126) | Prednisolone Drops 1% (Standard of Care) (N=55)
Intraocular pressure increased (Investigations) | 14 | 2
Iritis (Eye disorders) | 8 | 0
Headache (Nervous system disorders) | 1 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No